CLINICAL TRIAL: NCT00327262
Title: Multicenter, Phase III Study Comparing Imatinib (STI571, Glivec®) Standard Dose (400 Mg/Day) With Imatinib High Dose Induction (800 Mg/Day) Followed by Standard Dose Maintenance (400 Mg/Day) in Pretreated CML Patients in Chronic Phase
Brief Title: Comparing Imatinib Standard Dose With Imatinib High Dose Induction in Pretreated Chronic Myeloid Leukemia (CML) Patients in Chronic Phase
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central European Leukemia Study Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571AAT06
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2006-06-20 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Myeloid Leukemia
Keywords: chronic myeloid leukemia; Ph+; bcr/abl+; imatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib

SUMMARY:
This study will investigate the efficacy and tolerability of a short (6 months) high dose therapy followed by a standard dose compared to a continuous treatment with a standard dose of imatinib (Glivec®) in pretreated Philadelphia chromosome- positive (Ph+)/BCR-ABL+ CML patients in chronic phase.

DETAILED DESCRIPTION:
Patients with CML not achieving or losing a major cytogenetic response on whatever palliative treatment for CML, are at high risk to progress to accelerated phase and blast crisis. A new promising treatment with Imatinib (Glivec®), a tyrosine-kinase inhibitor, has been introduced recently. High rates of hematologic and cytogenetic responses can be achieved with Imatinib (Glivec®) at > = 300 mg/day in chronic phase CML patients that are refractory, resistant or intolerant to interferon-alpha. However, about 10 - 20% of these high risk patients will lose their response to Imatinib (Glivec®) within 1-2 years. Therefore, improvement of the treatment is warranted.

Since cytogenetic response rate is correlated to survival and the resistance to Imatinib (Glivec®) might be caused by mutations in the receptor, a more rapid decrease could lead to longer survival and/or less resistance development. In the initial 6 months of treatment, monotherapy with Imatinib (Glivec®) with a dose of 800 mg/day (high dose) should be more effective in the reduction of a high leukemic tumor burden, thereby allowing the residual normal progenitor and stem cells to expand. In addition, high dose Imatinib (Glivec®) should further improve the induction of a molecular response, as determined by quantitative reverse transcription polymerase chain reaction (RT-PCR), reducing the risk of relapse from residual malignant BCR-ABL positive cells.

This study will investigate the efficacy and tolerability of a short (6 months) high dose therapy followed by a standard dose compared to a continuous treatment with a standard dose of Imatinib (Glivec®).

In addition, the dynamics of the molecular and cytogenetic response will be investigated. Finally, the study will investigate the effect of this induction-maintenance concept on time-to-progression (TTP).

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years of age
2. BCR-ABL positive CML patients in chronic phase, confirmed by karyotype (Ph+) or RT-PCR.
3. Patients pretreated with any drug that is known to control the disease of CML in chronic phase except imatinib (Glivec®).
4. Patients without a major cytogenetic response at study entry (> 35% Ph+ metaphases in bone marrow cytogenetic analysis performed < 3 months before study entry).
5. Patients either intolerant to interferon-alpha (non-hematologic toxicity grade 3-4 for more than 2 weeks) or having received pretreatment for CML at least 12 months before study entry.
6. World Health Organization (WHO) status 0-2
7. Adequate end organ function, defined as the following:

   * total bilirubin < 1.5 x upper limit of normal (ULN)
   * SGOT and SGPT < 2.5 x ULN
   * creatinine < 1.5 x ULN
   * absolute neutrophil count (ANC) > 1.5 x 10 ^ 9/L
   * platelets > 100 x 10 ^ 9/L
8. Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
9. Written voluntary informed consent.

Exclusion Criteria:

1. Patients eligible for allogeneic bone marrow transplantation.
2. Patients in accelerated phase or blast crisis.
3. Known tuberculosis or other uncontrolled infection.
4. Other primary tumor of a different histological origin than the study indication (unless the relapse-free interval is > 5 years, and with the exception of cervical carcinoma in situ [CIS], basal cell epithelioma, or squamous cell carcinoma of the skin).
5. Major surgery within the last 14 days.
6. Known to be HIV positive.
7. Unstable medical disorder (except for indication) that excludes the patient in the opinion of the investigator.
8. Patient has received any other investigational agents within 28 days of first day of study drug dosing.
9. Patients with a WHO performance status score > 3
10. Patients with Grade III/IV cardiac problems as defined by the New York Heart Association criteria (i.e., congestive heart failure, myocardial infarction within 6 months of study).
11. Female patients who are pregnant or breast-feeding.
12. Refusal by female patients of childbearing age to use a safe contraceptive.
13. Patients with known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
14. Patients with any significant history of non-compliance to medical regimens or an inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2004-01; Study Completion 2008-12

PRIMARY OUTCOMES:
To determine the efficacy regarding major cytogenetic response within 12 months after randomization

SECONDARY OUTCOMES:
To determine the major cytogenetic response after 3 months versus 6-12 months after randomization
To determine the efficacy of the molecular response within 12 and 24 months after randomization
To determine the time to molecular progression within 24 months
To determine the dynamics of the molecular response within 3 and 6 months after randomization expressed as the slope decreases in BCR-ABL-transcripts
To determine tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Gastl, MD, Study Chair — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

REFERENCES:
- [Background] Talpaz M. Interferon-alfa-based treatment of chronic myeloid leukemia and implications of signal transduction inhibition. Semin Hematol. 2001 Jul;38(3 Suppl 8):22-7. doi: 10.1016/s0037-1963(01)90114-3. PMID 11526598
- [Background] O'Brien SG, Guilhot F, Larson RA, Gathmann I, Baccarani M, Cervantes F, Cornelissen JJ, Fischer T, Hochhaus A, Hughes T, Lechner K, Nielsen JL, Rousselot P, Reiffers J, Saglio G, Shepherd J, Simonsson B, Gratwohl A, Goldman JM, Kantarjian H, Taylor K, Verhoef G, Bolton AE, Capdeville R, Druker BJ; IRIS Investigators. Imatinib compared with interferon and low-dose cytarabine for newly diagnosed chronic-phase chronic myeloid leukemia. N Engl J Med. 2003 Mar 13;348(11):994-1004. doi: 10.1056/NEJMoa022457. PMID 12637609
- [Background] Kantarjian H, Talpaz M, O'Brien S, Garcia-Manero G, Verstovsek S, Giles F, Rios MB, Shan J, Letvak L, Thomas D, Faderl S, Ferrajoli A, Cortes J. High-dose imatinib mesylate therapy in newly diagnosed Philadelphia chromosome-positive chronic phase chronic myeloid leukemia. Blood. 2004 Apr 15;103(8):2873-8. doi: 10.1182/blood-2003-11-3800. Epub 2003 Dec 24. PMID 15070658
- [Background] Cortes J, Giles F, O'Brien S, Thomas D, Garcia-Manero G, Rios MB, Faderl S, Verstovsek S, Ferrajoli A, Freireich EJ, Talpaz M, Kantarjian H. Result of high-dose imatinib mesylate in patients with Philadelphia chromosome-positive chronic myeloid leukemia after failure of interferon-alpha. Blood. 2003 Jul 1;102(1):83-6. doi: 10.1182/blood-2003-01-0025. Epub 2003 Mar 13. PMID 12637317
- [Background] Sawyers CL, Hochhaus A, Feldman E, Goldman JM, Miller CB, Ottmann OG, Schiffer CA, Talpaz M, Guilhot F, Deininger MW, Fischer T, O'Brien SG, Stone RM, Gambacorti-Passerini CB, Russell NH, Reiffers JJ, Shea TC, Chapuis B, Coutre S, Tura S, Morra E, Larson RA, Saven A, Peschel C, Gratwohl A, Mandelli F, Ben-Am M, Gathmann I, Capdeville R, Paquette RL, Druker BJ. Imatinib induces hematologic and cytogenetic responses in patients with chronic myelogenous leukemia in myeloid blast crisis: results of a phase II study. Blood. 2002 May 15;99(10):3530-9. doi: 10.1182/blood.v99.10.3530. PMID 11986204
- [Background] Talpaz M, Silver RT, Druker BJ, Goldman JM, Gambacorti-Passerini C, Guilhot F, Schiffer CA, Fischer T, Deininger MW, Lennard AL, Hochhaus A, Ottmann OG, Gratwohl A, Baccarani M, Stone R, Tura S, Mahon FX, Fernandes-Reese S, Gathmann I, Capdeville R, Kantarjian HM, Sawyers CL. Imatinib induces durable hematologic and cytogenetic responses in patients with accelerated phase chronic myeloid leukemia: results of a phase 2 study. Blood. 2002 Mar 15;99(6):1928-37. doi: 10.1182/blood.v99.6.1928. PMID 11877262
- [Background] Kantarjian H, Sawyers C, Hochhaus A, Guilhot F, Schiffer C, Gambacorti-Passerini C, Niederwieser D, Resta D, Capdeville R, Zoellner U, Talpaz M, Druker B, Goldman J, O'Brien SG, Russell N, Fischer T, Ottmann O, Cony-Makhoul P, Facon T, Stone R, Miller C, Tallman M, Brown R, Schuster M, Loughran T, Gratwohl A, Mandelli F, Saglio G, Lazzarino M, Russo D, Baccarani M, Morra E; International STI571 CML Study Group. Hematologic and cytogenetic responses to imatinib mesylate in chronic myelogenous leukemia. N Engl J Med. 2002 Feb 28;346(9):645-52. doi: 10.1056/NEJMoa011573. PMID 11870241
- [Background] Druker BJ, Sawyers CL, Kantarjian H, Resta DJ, Reese SF, Ford JM, Capdeville R, Talpaz M. Activity of a specific inhibitor of the BCR-ABL tyrosine kinase in the blast crisis of chronic myeloid leukemia and acute lymphoblastic leukemia with the Philadelphia chromosome. N Engl J Med. 2001 Apr 5;344(14):1038-42. doi: 10.1056/NEJM200104053441402. PMID 11287973
- [Derived] Petzer AL, Fong D, Lion T, Dyagil I, Masliak Z, Bogdanovic A, Griskevicius L, Lejniece S, Goranov S, Gercheva L, Stojanovic A, Peytchev D, Tzvetkov N, Griniute R, Stanchev A, Grubinger T, Kwakkelstein M, Schuld P, Gastl G, Wolf D. High-dose imatinib induction followed by standard-dose maintenance in pre-treated chronic phase chronic myeloid leukemia patients--final analysis of a randomized, multicenter, phase III trial. Haematologica. 2012 Oct;97(10):1562-9. doi: 10.3324/haematol.2011.060087. Epub 2012 Apr 17. PMID 22511495
- [Derived] Petzer AL, Wolf D, Fong D, Lion T, Dyagil I, Masliak Z, Bogdanovic A, Griskevicius L, Lejniece S, Goranov S, Gercheva L, Stojanovic A, Peytchev D, Tzvetkov N, Griniute R, Oucheva R, Ulmer H, Kwakkelstein M, Rancati F, Gastl G. High-dose imatinib improves cytogenetic and molecular remissions in patients with pretreated Philadelphia-positive, BCR-ABL-positive chronic phase chronic myeloid leukemia: first results from the randomized CELSG phase III CML 11 "ISTAHIT" study. Haematologica. 2010 Jun;95(6):908-13. doi: 10.3324/haematol.2009.013979. Epub 2010 Feb 9. PMID 20145273